CLINICAL TRIAL: NCT06981650
Title: Video Education to Improve First Time Colonoscopy Outcomes: A Prospective Randomized Control Trial.
Brief Title: Video Education to Improve First Time Colonoscopy Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, John Trillo, Director of Gastroenetrology, South Brooklyn Health, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MED2024-555
Record Dates: First submitted 2025-04-24; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Colonoscopy Education
Keywords: colonoscopy
MeSH Terms: interventions — Videotape Recording; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- education (Active Comparator): standard education
  Interventions: Behavioral: education
- education plus video education (Experimental): standard education plus an additional approach
  Interventions: Behavioral: video; Behavioral: education

INTERVENTIONS:
Behavioral: video — use of a video
  Arms: education plus video education
Behavioral: education — standard talk and paper handout

SUMMARY:
The investigators compare video education plus standard education versus standard education for bowel preparation before a colonoscopy. The primary outcome will be the quality of bowel preparation.

DETAILED DESCRIPTION:
The investigators compare video education plus standard education versus standard education for bowel preparation before a colonoscopy and include a number of languages including English, Spanish, Russian, Haitian Creole, and Urdu. The educational content also includes psychological content based upon the Theory of Planned Behavior. The primary outcome will be the quality of bowel preparation, as measured by the Boston Bowel Preparation Scale (BBPS) score,

ELIGIBILITY:
Inclusion Criteria: all outpatients aged 18 to 75 years scheduled for their first screening colonoscopy

-

Exclusion Criteria: ● Contraindications for colonoscopy

* History of bowel surgery, particularly colorectal surgery
* Severe comorbid conditions (e.g., impaired hepatic, renal or bone marrow function, congestive heart failure, recent coronary artery disease)
* Chronic constipation (typically <3 bowel movements per week with hard stools, a feeling of incomplete evacuation, or abdominal discomfort) requiring the use of laxatives
* Pregnancy or lactation
* Prisoners
* Diagnosis of inflammatory bowel disease
* Inability to use video presentation devices (e.g., blindness)
* Active cancers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale (continuous) | Perioperative/Periprocedural
  Quality of bowel preparation measured by the Boston Bowel Preparation Scale. Scores range from 0 through 3. Higher scores indicate a better outcome..

SECONDARY OUTCOMES:
Boston Bowel Preparation Scale (categorical) | Perioperative/Periprocedural
  Boston Bowel Preparation Scale adequacy of preparation score ≥ 2 in all regions.
  Quality measured by the Boston Bowel Preparation Scale. Scores range from 0 through 3. Higher scores indicate a better outcome..
Polyp detection rate proportion | Perioperative/Periprocedural
  Proportion of individuals undergoing a colonoscopy in whom at least one polyp is detected. Values range from 0 through 1. Higher values indicate a better outcome.
Adenoma detection rate proportion | Perioperative/Periprocedural
  Proportion of individuals undergoing a colonoscopy in whom at least one adenomatous polyp is found. Values range from 0 through 1. Higher values indicate a better outcome.
Cecal intubation rate proportion | Perioperative/Periprocedural
  Proportion of colonoscopies in which the endoscope successfully reaches the caecum. Values range from 0 through 1. Higher values indicate a better outcome.
Withdrawal time | Perioperative/Periprocedural
  Duration in minutes taken to withdraw the colonoscope from the caecum to the rectum. Values range from 1 through 60. Higher values indicate a worse outcome.
Adherence to bowel preparation instructions | Perioperative/Periprocedural
  Following what was told to do by bowel preparation instructions. Total of 7 original questions scored as no for 0 or yes for 1 with a total score ranging from 0 through 7. Higher values indicate a better outcome.
Amsterdam Preoperative Anxiety and Information Scale | baseline
  Self-assessed at baseline using the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Scores range from 6 through 30. Higher scores greater anxiety.
Overall experience with the bowel preparation process | Perioperative/Periprocedural
  Self-report about experience with the bowel preparation process. One original question with 5 choices of very unpleasant, unpleasant , neutral , pleasant , very pleasant . There is no score. The best answer would be "very pleasant."
Desire to undergo future colonoscopies if indicated | Perioperative/Periprocedural
  Self-report about having another colonoscopy. One original question with 5 choices of strongly disagree, disagree, neutral, agree , strongly agree. The best answer would be "strongly agree."

IPD SHARING:
Plan to Share IPD: Yes
Deidentfied data based upon a reasonable request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study using data is published.
Access Criteria: Academic researchers

REFERENCES:
- [Background] Mahmood S, Farooqui SM, Madhoun MF. Predictors of inadequate bowel preparation for colonoscopy: a systematic review and meta-analysis. Eur J Gastroenterol Hepatol. 2018 Aug;30(8):819-826. doi: 10.1097/MEG.0000000000001175. PMID 29847488